CLINICAL TRIAL: NCT00794430
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre, Parallel Group Study of the Safety, Tolerability and Efficacy of V3381 for up to 13 Weeks in Patients With Diabetic Peripheral Neuropathic Pain (DPNP)
Brief Title: Study of the Safety, Tolerability and Efficacy of V3381 in Patients With Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V3381-2DPNP-02
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2015-01

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Safety; Tolerability; Efficacy; Patients; Diabetic peripheral neuropathic pain.
MeSH Terms: interventions — indantadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V3381 (Experimental): V3381: titrated from 100 mg bid to maximum 400 mg bid over 4 weeks followed by maintenance phase at highest tolerated dose. Total duration of treatment 13 weeks.
  Interventions: Drug: V3381
- Placebo (Placebo Comparator): Placebo to match V3381, 100 mg, given according to the same regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V3381 — 100 mg capsules, titrated to a maximum of 400 mg bid for 13 weeks
  Other Names: Indantadol
  Arms: V3381
Drug: Placebo — Capsule, bid, for 13 weeks
  Arms: Placebo

SUMMARY:
Randomised, double-blind, placebo-controlled, parallel group, multicentre study of oral doses of V3381, titrated to effect. A 2-week single-blind run-in period will be followed by a 13 week double-blind titration and maintenance phase. Doses will be titrated up in 100 mg bid increments every one or two weeks, starting from 100 mg bid. A 2 week follow-up period will conclude patient participation in the study.

DETAILED DESCRIPTION:
Patients who provide written informed consent will be screened for entry into the study.

Patients will initially enter a 2-week single-blind run-in phase, during which they will complete an 11 point numerical pain rating scale (NPRS) on their average daily pain; patients with a mean weekly score of >4 and <9 will be allowed to continue in the study to randomisation (unless they have exhibited a >50% decrease in pain score, compared to the Day -14 score, during the run-in).

Patients will be randomised to receive either Placebo (PL) bid (n=75) or V3381 (n=75) and will initially be treated with 100 mg V3381 (or placebo equivalent) twice daily (bid) for one week. Patients will remain on the same study treatment throughout the trial. At the end of one week those patients who adequately tolerated study medication will escalate the dose of V3381 to 200 mg bid on a blinded basis. Patients who do not tolerate 100 mg bid will be withdrawn.

After one week of treatment at the 200 mg bid dose level, those subjects who continue to tolerate adequately 200 mg bid study drug will escalate to 300 mg bid. Subjects who have not tolerated the 200 mg bid dose may revert to the 100 mg bid dose and should remain at this dose level for the remainder of the trial.

After a further 2 weeks of treatment those subjects who continue to tolerate adequately 300 mg bid study drug will escalate to 400 mg bid. Subjects who have not tolerated the 300 mg bid dose may revert to the 200 mg bid dose and should remain at this dose level for the remainder of the trial.

Subjects will then remain on these doses (that is, the dose of V3381 or placebo which they tolerate) for the remaining 9 weeks of the treatment period. In exceptional cases of new intolerability developing, patients may be down-titrated to the next lower dose level.

All patients will be provided with the rescue medication paracetamol (acetaminophen) 650 mg up to four times daily (North America [NA]) or 1000 mg up to three times daily (Europe [EU]) to supplement study drug, should they wish to do so, throughout the study, including the single-blind placebo phase.

Patients will be expected to attend the clinic 9 times (at Screening, Baseline, Week 1, Week 2, Week 4, Week 7, Week 10, Week 13 and Follow-up clinic visits) for safety and efficacy assessments. The safety assessments will include biochemistry, haematology and urinalysis tests, 12 lead electrocardiogram (ECG), vital signs, recording of adverse events, Beck Depression Inventory, review of medication compliance, and of blood glucose control.

The following assessments will also be conducted at each clinic visit during treatment and follow up:

* Modified Brief Pain Inventory for diabetic painful neuropathy (DPN)
* Neuropathic Pain Symptom Inventory
* Patient Clinical Global Impression score
* Investigator Clinical Global Impression score

The Medical Outcomes Survey Short Form-36, Version 2 will be assessed at baseline and Visit 8.

Subjects will complete home diaries on a daily basis on which they will rate average pain using the 11-point Likert NPRS. Sleep interference scores, worst daily pain and use of rescue medication will also be recorded on the daily diaries.

A Steering Committee will be established to provide oversight of the conduct of the trial. A Data Safety Monitoring Board (DSMB) will be convened to periodically review patient safety.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female aged 18 - 75 (18-65 Czech Republic)
3. Diagnosis of diabetes mellitus
4. No change in diabetes medications within 4 weeks before screening
5. Daily pain attributed to diabetic neuropathy present for at least 6 months immediately prior to study entry
6. Presents with pain due to bilateral peripheral neuropathy caused by Type I or Type II diabetes mellitus. Pain must have begun in the feet, with relatively symmetrical onset. Diagnosis confirmed by a score of at least 2 on Section B of the MNSI
7. Judged to be reliable and agree to keep all appointments required by the protocol
8. Females should be of non child-bearing potential (i.e. surgically sterilized or >1 year post-menopause). Male subjects who are sexually active with a female partner of child bearing potential must agree to use a barrier method of contraception (eg condom, diaphragm or cervical cap in the female female partner) for the duration of the study (until the follow up visit)

   Additionally, at the baseline visit:
9. A mean average pain intensity of at least 4, but less than or equal to 9, on an 11 point Likert NPRS recorded twice daily during the two week placebo run-in; any patient who experiences a >30% decrease in the mean pain score compared to Day -14 during placebo run-in will be excluded, regardless of whether their final score is >4
10. Full completion of daily diaries for at least 11 of the days up to Day -1
11. Compliance in taking placebo run-in medication twice daily for at least 11 of the days up to Day -1

Exclusion Criteria:

1. Any clinically significant neurologic disorders (except DPNP)
2. Any clinically significant or unstable medical or psychiatric condition that would affect the patient's ability to participate in the study
3. Prior renal transplant, current renal dialysis
4. Pernicious anemia
5. Untreated hypothyroidism
6. Amputations or persistent ulceration due to diabetes mellitus
7. Any cardiovascular condition that would contraindicate the use of sympathomimetic amines
8. Uncontrolled hypertension
9. Known or at high risk of HIV infection
10. Any anticipated need for surgery during the study
11. Increased risk of seizures (defined as a history of seizure disorder (including alcoholic seizures), family history of seizures and history of head trauma that resulted in loss of consciousness or concussion).
12. Any malignancy in the past 2 years (except basal cell carcinoma)
13. Pain that cannot be clearly differentiated from, or conditions that interfere with, the assessment of diabetic neuropathic pain
14. Use of anticonvulsants, antidepressants (particularly MAO inhibitors), or prescription membrane-stabilizing agents, including topical therapies. Patients currently taking drugs in these classes may have them discontinued prior to entry into the placebo run-in period.
15. Use of opioids, especially meperidine (pethidine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of V3381 in patients with diabetic neuropathic pain at doses of up to 400 mg bid | 17 weeks

SECONDARY OUTCOMES:
Determine the efficacy of V3381 in the treatment of diabetic peripheral neuropathic pain at does of up to 400 mg bid | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sang, Principal Investigator — Brigham and Women's Hospital
Locations (31):
- United States (9):
  - Clinical Trials Inc, Little Rock, Arkansas
  - Renstar Inc, Ocala, Florida
  - Radiant Research Inc, St. Petersburg, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Radiant Research Inc, Cincinnati, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - dgd Research, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
- Canada (2):
  - LMC Endocrinology, Thornhill
  - LMC Endocrinology, Toronto
- Czechia (10):
  - Private Clinic, Brno, Brno
  - Nemocnice Ceske Budejovice, České Budějovice, Ceske Budejovice
  - Private Clinic, Holešov, Holesov
  - Private Clinic, Hranice, Hranice
  - Smetanovy sady, Karlovy Vary, Karlovy Vary
  - Neurologicke oddeleni, Pardubice, Pardubice
  - Private Clinic, Michnova 1622/4, Prague, Prague
  - ResTrial s.r.o., Prague, Prague
  - Lekarsky dum Ormiga, Zlín, Zlín
  - Diabetology Center, Zlín
- United Kingdom (10):
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Ipswich Hospital NHS Trust, Ipswich, Suffolk
  - Barnsley Hospital, Barnsley
  - MAC UK Neuroscience, Blackpool
  - Addenbrookes Hospital, Cambridge
  - Colchester Hospital University NHS Foundation Trust, Colchester
  - Pallium Research Group (Seacroft Hospital), Leeds
  - St John's Hospital, Livingston
  - Barts and The London NHS Trust, London
  - Royal Hallamshire Hospital, Sheffield